CLINICAL TRIAL: NCT00646295
Title: Pascal Dynamic Contour Tonometer Intraocular Pressure and Ocular Pulse Amplitude in Patients With Thyroid Related Orbitopathy: A Comparison to Goldmann Tonometer and to Muscles Characteristics on Orbital CT Scan
Brief Title: Pascal Pascal Dynamic Contour Tonometer (DCT) Intraocular Pressure and Ocular Pulse Amplitude in Patients With Thyroid Related Orbitopathy: A Comparison to Goldmann Tonometer and to Muscles Characteristics on CT Scan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ehud Rechtman,/MD & Guy Ben Simon/MD, Goldschleger Eye Institute, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-08-5058-ER-CTIL
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Thyroid Related Orbitopathy
Keywords: TRO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): To measure the IOP (with Goldmann and Pascal DCT tonometers) and OPA (with Pascal DCT) in primary and upright gazes
  Interventions: Device: To measure the IOP (with Goldmann and Pascal DCT tonometers) and OPA (with Pascal DCT) in primary and upright gazes

INTERVENTIONS:
Device: To measure the IOP (with Goldmann and Pascal DCT tonometers) and OPA (with Pascal DCT) in primary and upright gazes — Pascal Dynamic Contour Tonometer Goldmann Applanation Tonometer
  Other Names: Pascal Dynamic Contour Tonometer; Pascal DCT; Goldmann tonometer

SUMMARY:
Thyroid related orbitopathy (TRO) is an autoimmune disease. Clinical features include: orbital pressure pain, ocular soft tissue swelling, muscle enlargement around the eyeball, eyelid retraction and bulging of the eye anteriorly out of the orbit. In many cases, the cornea may become too dry, and as a result, corneal ulcers may form, which can become infected. In severe cases, damage to the optic nerve can occur secondary to optic nerve compression by enlarged muscles in the orbit.

Inflammation with soft tissue swelling occurs in the 1st stage of the disease. Scar formation can occur in the 2nd phase. The muscles under and nasal to the eyeball are most commonly involved. In many patients, intra-ocular pressure (IOP) can increase in primary. IOP in upgaze (when looking up) can increase.

Goldmann applanation is the standard device to measure the IOP. It measures the average IOP (between the "systolic", when the heart contracts, to the diastolic IOP, when the heart relaxes). Pascal Dynamic Contour Tonometer is a new device that can measure IOP and ocular pulse amplitude (OPA) which is the difference between diastolic IOP and systolic IOP. The choroid is a vascular layer inside the eyeball that feeds part of the retina (the retina is like the film in a non-digital camera). OPA is suggestive of choroidal blood flow. IOP measurements using Pascal Dynamic Contour Tonometer are less influenced by corneal thickness as opposed to Goldmann applanation which measures higher values in thicker corneas. In the current study we are interested in measuring the relationships between measurements taken with Goldmann applanation (IOP) and those taken with the Pascal Dynamic Contour Tonometer (IOP and OPA). In addition, we will investigate the effect of orbital muscle enlargement on IOP/OPA following an up gaze position (looking up).

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 yr
2. agree to participate in the study and willing to sign an informed consent

Exclusion Criteria:

1. other ocular diseases (besides cataract and mild hypertensive retinopathy)
2. previous history of eye surgery besides cataract extraction and Nd:YAG laser capsulotomy
3. moderate to severe cataract that precludes fundus examination
4. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
IOP in primary and upright gazes measured by Goldmann and Pascal Dynamic Contour tonometers. | one visit

SECONDARY OUTCOMES:
The change in IOP & OPA as measured by Pascal Dynamic Contour Tonometer following an upright gaze | one time

CONTACTS AND LOCATIONS:
Locations (1):
- Goldschleger Eye Institute, Sheba Medical Center, Tel-Hashomer, Ramat-Gan, Israel